CLINICAL TRIAL: NCT02950454
Title: The Effect of High Intensity Interval Training on Cardiovascular Fitness in People With Progressive Multiple Sclerosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Ayrshire and Arran (Other); AKM (Other)
Responsible Party: Principal Investigator, Evan Campbell, PhD Student, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Multiple Sclerosis, Progressive
Keywords: Progressive Multiple Sclerosis; Rehabilitation; Exercise
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 8 weeks of twice weekly high intensity interval training. Session protocol: 2 minute warm up at nominal resistance on cycle ergometer, 6 six intervals of 80-95% heart rate max interspersed with 6 intervals of 1.5 minute working rest. Then 3 minutes cool down.
  Interventions: Other: High intensity interval training
- control (Active Comparator): 8 weeks of twice weekly continuous moderate intensity exercise. Session protocol: 2 minutes warm up at nominal resistance on cycle ergometer, 20 minutes at 60-70% heart rate max. Then 3 minutes cool down.
  Interventions: Other: Continuous moderate exercise

INTERVENTIONS:
Other: High intensity interval training — 1.5 min intervals at 80-95% heart rate max on cycle ergometer 1.5 min intervals at nominal resistance on cycle ergometer
  Arms: Intervention
Other: Continuous moderate exercise — 20 min at 60-70% heart rate max on cycle ergometer
  Arms: control

SUMMARY:
This is a pilot trial to explore the cardiovascular of eight weeks of twice weekly high intensity interval training in people with progressive multiple sclerosis. A control group of people with progressive multiple sclerosis will undergo continuous moderate intensity exercise, twice weekly for 8 weeks.

DETAILED DESCRIPTION:
This is a pilot trial to explore the cardiovascular of eight weeks of twice weekly high intensity interval training in people with progressive multiple sclerosis. A control group of people with progressive multiple sclerosis will undergo continuous moderate intensity exercise, twice weekly for 8 weeks.

The training program will entail 6x1.5 minute intervals working at 80-95% heart rate max on a cycle ergometer. Each interval will be interspersed with 1.5 minutes of working rest at a light resistance of the participant's choosing.

The continuous moderate intensity exercise program will entail 20 minutes on a cycle ergometer working at 60-70% heart rate max.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a progressive form of MS
* Aged 18 years or older
* Known to members of staff of the MS service NHS Ayrshire & Arran
* Ability to attend Douglas Grant Rehabilitation centre twice a week for eight weeks
* EDSS 4-6.0
* Able to cycle on ergometer

Exclusion Criteria:

* A relapse of symptoms requiring treatment within the past three months.
* A respiratory condition that would be exacerbated by high intensity exercise including but not limited to: chronic obstructive pulmonary disorder, uncontrolled or poorly controlled asthma.
* Uncontrolled high pressure at screening (>190/100 mmHg)
* Cognitive impairment affecting ability to understand instructions as noted in patient's notes.
* Currently engaging in another research trial for their MS or that may affect their physiological or cardiovascular outcomes
* Weighing more than 110 kg (weight limit of ergometer)
* Any pathology or medical intervention that would preclude high intensity exercise, maximal exertion testing or could attenuate the cardiovascular effect of exercise including but not limited to: unstable angina; diabetes; peripheral vascular disease or intermittent claudication; having a pace maker or medicine pump; surgical clips; having another neurological condition other than MS; and pregnancy. To be established from patient's notes and at screening session.
* A serious cardiovascular event in the past year including but not limited to: transient ischaemic attack, cerebrovascular event and myocardial infarction.
* Taking any of the following medication: beta blockers; vasodilators; ACE inhibitors; diuretics or any other medication that could cause exercise induced hypotension; hypoglycaemic insulin; metformin or other oral insulin medicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
heart rate max | 8 weeks
  Maximal heart rate elicited during a maximal exertion test

SECONDARY OUTCOMES:
Resting blood pressure | 8 weeks
Resting heart rate | 8 weeks
Brain derived neurotrophic factor | 8 weeks
  Hormone important for brain growth and protection
Lactate | 8 weeks
  Waste materials from exercise in blood
Lipoprotein profile | 8 weeks
  Indication of how much good and how much bad cholesterol is in blood
MSIS-29 version 2 | 8 weeks
  Questionnaire giving physical and psychological impact of MS
Hospital anxiety and depression scale | 8 weeks
  Questionnaire giving a score of depression and anxiety
Timed 25 foot walk test | 8 weeks
  Measure of walking speed
Symbol digit modalities test | 8 weeks
  Measure of mental processing speed
Fatigue severity scale | 8 weeks
  Questionnaire which gives measure of fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No